CLINICAL TRIAL: NCT04768231
Title: Safety of Rifampicin at High Dose for the Treatment of Adult Subjects With Complex Drug Susceptible Pulmonary and Extrapulmonary Tuberculosis
Brief Title: Rifampicin at High Dose for Difficult-to-Treat Tuberculosis
Acronym: RIAlta
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: University Medical Center Groningen (Other); Radboud University Medical Center (Other); Centro Hospitalar De São João, E.P.E. (Other); Instituto Nacional de Enfermedades Respiratorias y del Ambiente, Paraguay (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIAlta-1; 2020-003146-36 (EudraCT Number)
Record Dates: First submitted 2021-02-15; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis
Keywords: Rifampicin; Tuberculosis; Safety
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Single intervention group compared with historical controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- R35HZE (Experimental): Participants treated with rifampicin at a dose of 35 mg per kilogram of body weight per day, added to the standard doses of isoniazid, pyrazinamide and ethambutol.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Rifampin — The target dose of 35mg/kg will be reached supplementing fixed-dose combination tablets (standard dose) with rifampin-only tablets.
  Other Names: Rifampicin

SUMMARY:
The purpose of this study is to assess the safety of rifampicin given at a dose three times as the standard one, in persons with tuberculosis that belong to groups that have not been widely included in previous trials.

DETAILED DESCRIPTION:
A prospective, one-arm, open-label trial to evaluate the safety of rifampicin at 35mg/kg per day, added to the remaining standard first-line drugs, in subjects with tuberculosis belonging to groups that have been underrepresented in previous trials: persons living with HIV, older than 65 years, malnourished, diabetics, and chronic stable liver disease. The main outcome is the rate of severe adverse events and adverse events leading to treatment modification as compared to that in a historical cohort (patietns belonging to these groups treated in the same centers from 2017-2019). Microbiological efficacy and extended follow-up data until one year after treatment will also be collected.

ELIGIBILITY:
Inclusion criteria:

The participant must fulfill either criteria nr. 1-4 AND nr. 5 OR criteria nr. 1-4 AND 6, AND anyone of 7-14:

1. Subjects with confirmed or probable pulmonary or extra pulmonary DS-TB.
2. Informed consent provided.
3. Positive smear, positive Xpert® MTB/RIF test, positive M. tuberculosis culture (confirmed cases) OR histological study compatible with necrotizing granulomas OR a liquid biochemistry (pleural, pericardial, ascites or cerebrospinal fluid) suggestive of TB together with clinical symptoms resembling TB disease in the absence of any other possible cause (probable cases).
4. Female participants of childbearing age must have a negative pregnancy test at baseline.

   AND
5. Age ≥ 60 years old. OR
6. Age ≥ 18 years AND one of the following
7. Body mass index ≤ 18.5
8. Human Immunodeficiency Virus (HIV) infection.
9. Diabetes Mellitus
10. Hepatitis C virus (HCV) infection (positive HCV serology)
11. Hepatitis B virus (HBV) infection (positive HBV surface antigen or anti-core antibodies)
12. Daily alcohol intake ≥ 2 units of alcohol (1 unit of alcohol: 4% alcohol 250ml (ie beer); 4.5% alcohol 218ml (i.e. cider); 13% alcohol 76ml (i.e. wine); 40% alcohol 25ml (i.e. whisky))
13. Chronic liver disease of any other cause (metabolic, toxic, autoimmune)
14. Central Nervous System TB involvement

Exclusion criteria:

Subjects will be excluded from entry if ANY ONE of the criteria listed below is met:

1. Rifampicin resistance confirmation.
2. Barthel index <40 for subjects older than 60 years old.
3. Signs of significant liver disease:

   * Liver enzymes (AST or ALT) > 5x upper limit of normal
   * Total bilirubin > 3x upper limit of normal
   * Subjects with a Child-Pugh grade C cirrhosis or acute decompensation of their chronic liver disease at enrolment.
   * Any other grade 3-4 hepatobiliary alteration according to the CTCAE v5.
4. Subjects with known allergy or sensitivity to rifampicin, or any of the other components of DS-TB treatment.
5. Treatment with any of the following: rifampicin, isoniazid, pyrazinamide, ethambutol, levofloxacin, or moxifloxacin within the last month for at least 14 days or current TB treatment for more than 7 days.
6. The subject is enrolled in any other investigational trial that includes a drug intervention.
7. Subjects with solid organ transplantation or bone marrow transplantation.
8. Subjects with an active onco-hematological neoplasm requiring chemotherapy or immune therapy.
9. Previous severe pulmonary disease, other than pulmonary DS-TB, according to local investigator.
10. Pre-existing epilepsy or psychiatric disorder according to local investigator.
11. Ischemic heart disease OR severe arrhythmia within 6 months OR Atrial Fibrillation with oral anticoagulant therapy indication when transitioning to low-molecular weight heparin is not feasible.
12. Positive pregnancy test
13. Breastfeeding women.
14. The subject used any drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes which are involved in the degradation pathways of rifampicin within the time windows specified in table 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of rifampicin at 35mg/kg/day | During the first 8 weeks after treatment start
  Rate of grade 3 or higher adverse events as compared to that in historical controls

SECONDARY OUTCOMES:
Efficacy of rifampicin at 35mg/kg/day in pulmonary tuberculosis | At week 8 after treatment start
  Rate of sputum liquid culture conversion (only pulmonary TB participants)
Tolerability of rifampicin at 35mg/kg/day | During the first 8 weeks after treatment start
  Rate of adverse events of any grade as compared to that in historical controls

OTHER OUTCOMES:
Bactericidal activity in pulmonary tuberculosis | During the first 8 weeks after treatment start
  To describe the rate of sputum smear conversion, decline in bacterial load (measured as logCFU/mL), ant time-to-negative smear and culture.
Pharmacokinetics of rifampicin: Maximum concentration (Cmax) | After 4 weeks of treatment
  To describe the Camx of rifampicin at 35mg/kg in the population included in the study. A spare-sample strategy sill be used with blood samples taken at 2, 4, and 6 hours after rifampicin administration.
Pharmacokinetics of rifampicin: Time to maximum concentration (Tmax) | After 4 weeks of treatment
  To describe the Tmax of rifampicin at 35mg/kg in the population included in the study. A spare-sample strategy sill be used with blood samples taken at 2, 4, and 6 hours after rifampicin administration.
Pharmacokinetics of rifampicin: Area Under the Curve (AUC) 0-24 | After 4 weeks of treatment
  To describe the AUC0-24 of rifampicin at 35mg/kg in the population included in the study. A spare-sample strategy sill be used with blood samples taken at 2, 4, and 6 hours after rifampicin administration. The AUC 0-24h will be modelled accodring to the methods described in Magis-Escurrra et al, 2014.
Pharmacogenetics: analyze the variants in SLCO1B1, ABCB1, UGT1A, and PXR genes | After 4 weeks of treatment
  Analyze the polymorphisms in SLCO1B1, ABCB1, UGT1A, and PXR genes and their correlation with pharmacokinetic measures from previous outcomes.
Pharmacodynamics: correlate the AUC0-24/MIC ratio with culture conversion rate | After 4 weeks of treatment (AUC0-24/MIC) and 8 weeks (culture conversion rate)
  Correlate the pharmacokinetic measure AUC0-24 to the MIC (Minimum Inhibitory Concentration) ratio with the rate of culture conversion of sputum sample at 8 weeks in liquid culture medium.
AeoNose™ signature during treatment in pulmonary tuberculosis | Baseline and weeks 1, 2, 4, 6 and 8.
  Evaluate the response to treatment in the exhaled volatile particles signature by means of an electronic nose device: AeoNose™ (The eNose company, the Netherlands)
Correlation of AeoNose™ with the bactericidal activity in pulmonary tuberculosis | Baseline and weeks 1, 2, 4, 6 and 8.
  Correlation of the changes in signature by means of an AeoNose™ and the changes in bacillary load during the first 8 weeks of treatment and the culture conversion rate at 8 weeks.
Health Economics | During the 6-month standard treatment period.
  To describe tuberculosis associated costs and the incidence of catastrophic costs using the EUSAT-RCS questionnaire based on the WHO handbook for economic studies in tuberculosis in a subgroup of the participants.
Quality of life | During the 6-month standard treatment period.
  To describe the changes in quality of life during tuberculosis treatment using the SF-12 questionnaire and the St George's respiratory questionnaire (for pulmonary TB participants) of a subgroup of the included participants
Extended follow-up: safety | Up to 12 months after the end of TB treatment.
  After the end of the intervention (8 weeks) data will be collected about severe (grade 3 or higher) or serious adverse events.
Extended follow-up: cure, treatment failure, relapse | Up to 12 months after the end of TB treatment.
  After the end of the intervention (8 weeks) data will be collected about clinical outcomes as defined by the WHO (cure, treatment failure, relapse).

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Sánchez-Montalvá, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (5):
- Netherlands (2):
  - University Medical Center, Groningen
  - Radboud University Medical Center, Nijmegen
- Instituto Nacional de Enfermedades Respiratorias y del Ambiente, Asunción, Paraguay
- Centro Hospitalario Universitario de Sao Joao, Porto, Portugal
- Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upn request to the EUSAT-consortium Steering Committee
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the end of the study; without specified limit.

REFERENCES:
- [Background] van Ingen J, Aarnoutse RE, Donald PR, Diacon AH, Dawson R, Plemper van Balen G, Gillespie SH, Boeree MJ. Why Do We Use 600 mg of Rifampicin in Tuberculosis Treatment? Clin Infect Dis. 2011 May;52(9):e194-9. doi: 10.1093/cid/cir184. PMID 21467012
- [Background] Seijger C, Hoefsloot W, Bergsma-de Guchteneire I, Te Brake L, van Ingen J, Kuipers S, van Crevel R, Aarnoutse R, Boeree M, Magis-Escurra C. High-dose rifampicin in tuberculosis: Experiences from a Dutch tuberculosis centre. PLoS One. 2019 Mar 14;14(3):e0213718. doi: 10.1371/journal.pone.0213718. eCollection 2019. PMID 30870476
- [Background] Steingart KR, Jotblad S, Robsky K, Deck D, Hopewell PC, Huang D, Nahid P. Higher-dose rifampin for the treatment of pulmonary tuberculosis: a systematic review. Int J Tuberc Lung Dis. 2011 Mar;15(3):305-16. PMID 21333096
- [Background] Magis-Escurra C, Later-Nijland HM, Alffenaar JW, Broeders J, Burger DM, van Crevel R, Boeree MJ, Donders AR, van Altena R, van der Werf TS, Aarnoutse RE. Population pharmacokinetics and limited sampling strategy for first-line tuberculosis drugs and moxifloxacin. Int J Antimicrob Agents. 2014 Sep;44(3):229-34. doi: 10.1016/j.ijantimicag.2014.04.019. Epub 2014 Jun 9. PMID 24985091
- [Derived] Espinosa-Pereiro J, Ghimire S, Sturkenboom MGG, Alffenaar JC, Tavares M, Aguirre S, Battaglia A, Molinas G, Tortola T, Akkerman OW, Sanchez-Montalva A, Magis-Escurra C. Safety of Rifampicin at High Dose for Difficult-to-Treat Tuberculosis: Protocol for RIAlta Phase 2b/c Trial. Pharmaceutics. 2022 Dec 20;15(1):9. doi: 10.3390/pharmaceutics15010009. PMID 36678638
- See also: EUSAT consortium website — http://www.eusattb.net/